CLINICAL TRIAL: NCT06164691
Title: The Effect of Peri-surgery Blue and Amber Light Exposure in Subjects Undergoing Medical and Surgical Treatment of Cancer
Brief Title: Blue and Amber Light Exposure in Patients With Rectal and Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI terminated study due to lack of enrollment.
Sponsor: Matthew Neal MD (Other)
Responsible Party: Sponsor-Investigator, Matthew Neal MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY22060036
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Neoplasms; Rectal Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization will achieved with block randomization on the following characteristics:
  1. Type of cancer: group 1: pancreatic cancer; group 2: rectal cancer.
  2. Stage of cancer as defined by Tumor Node Metastasis classification.
  b. Age (<55 years, >/= 55 years)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Blue light (Experimental): This cohort will be exposed to bright (1700 lux) blue (peak 442 nm) light for 4 hours each morning for 3 days prior to and 3 days following each chemotherapy infusion.They will be exposed to bright (1700 lux) blue (peak 442 nm) light for 1 hour each morning during radiation treatments.
  Interventions: Device: Blue light
- Amber light (Experimental): This cohort will be exposed to bright (1700 lux) amber (peak 617 nm) light for 4 hours each morning for 3 days prior to and 3 days following each chemotherapy infusion.They will be exposed to bright (1700 lux) amber (peak 617 nm) light for 1 hour each morning during radiation treatments
  Interventions: Device: Amber light
- Ambient white light (Active Comparator): This cohort will be exposed to usual, ambient white lighting of the environment during chemotherapy and radiation treatments.
  Interventions: Other: Ambient White Light

INTERVENTIONS:
Device: Blue light — Participants undergoing this intervention will be exposed to blue (442nm) light.
  Arms: Blue light
Device: Amber light — Participants undergoing this intervention will be exposed to amber (617nm) light.
  Arms: Amber light
Other: Ambient White Light — This cohort will be exposed to usual, ambient white lighting of the environment during chemotherapy and radiation treatments
  Arms: Ambient white light

SUMMARY:
This study will evaluate light therapy used in combination with standard therapies for pancreatic and rectal cancer. Participants will receive chemotherapy, radiation, and surgical treatments identical to that they had not been involved in the study. The only alteration is that some participants will be exposed additionally to either blue or amber light using commercially available seasonal affective disorder (SAD) lights that are approved for human use. Participants will use the SAD light in their own homes throughout the course of their radiation and chemotherapy treatments. They will wear goggles that filter with the desired color of light. As a comparison, another group of participants will be exposed only to their usual lighting conditions. The assignment to blue light, amber light, or usual light groups will be random.

In addition to the light exposure, participants will be asked to have 10 mL of blood drawn for research purposes at 4 time points. This blood will be analyzed for markers of inflammation and circadian clock activation. Participants also will be asked to complete surveys at 3 time points. These surveys will evaluate for effects changs in sleep, pain, and quality of life. Finally, participants will be asked to wear a small clip-on light sensor and a heart rate variability monitor for 7 days. These monitors will provide information on the level of light exposure and the participant's physiologic response to the light. For participants going on to surgery, we will obtain a small sample of the resected pancreas or rectal tumor for research analysis. The investigators will obtain this sample only after the necessarily analysis has been performed for their clinical care.

DETAILED DESCRIPTION:
The investigators incorporate appropriate control participants, which include participants who are matched for stage and age and who undergo neoadjuvant chemoradiation and/or surgery but who are not exposed to modulation of their environmental light.

There are no deviations from the standard of care for these patients. They will be receiving care identical to that had they not been involved in this study. The only alteration is that some participants will be exposed additionally to either blue or amber light. The investigators use commercially available seasonal affective disorder (SAD) lights that are already approved for therapeutic human use. These lights are small and portable and approved for use for seasonal affective disorder (SAD). The investigators have used them in other human trials and have not identified any adverse or unexpected events.

The participants will be asked to have 10 mL of blood drawn for research purposes at 4 time points to assess for markers of the inflammatory response and circadian clock activation. Additionally, they will be asked to complete surveys at 3 time points to assess for quality-of-life measures. They will be asked to wear a small light sensor and a heart rate variability monitor for 7 days to measure the adequacy of light exposure and physiologic response to the exposure, respectively.

In the participants who undergo definitive operative resection (e.g., Whipple (pancreaticoduodenectomy) procedure, mesorectal proctectomy), we will analyze a sample of the resected specimen. The investigators will obtain this sample only after complete pathological examination and reporting in accordance with best practices of care. Thus, the sample being acquired for research purposes is discarded biological tissue and no additional sampling is performed. In fact, there are absolutely no deviations or interference with the processes of delivering care.

ELIGIBILITY:
Inclusion Criteria:

1. greater than 18 and less than 80 years of age
2. adenocarcinoma of the pancreas (unresectable) or adenocarcinoma of the rectum (stage II or III).

Exclusion Criteria:

1. Prior chemotherapy (inability to determine the integrity of the immune response)
2. Autoimmune disorder, immunosuppression therapy, or immunocompromised state (inability to determine the integrity of the immune response)
3. Blindness or other significant vision disorder or prior traumatic brain injury (the inability to determine the integrity of functional optic and suprachiasmatic pathways)
4. Hematological disease - e.g., myelodysplastic syndrome, leukemia (inability to determine the integrity of the immune response)
5. Bipolar disorder or schizophrenia (potential heightened symptoms)
6. Refusal/ineligible to undergo neoadjuvant chemotherapy and/or radiation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-08-14 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Neal, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification will be shared. A data dictionary will also be made available. Data will be available beginning 12 months and ending 36 months following article publication. Data will be shared with those researchers who provide a methodologically sound proposal. Only those data necessary to achieve the aims in the approved proposal will be shared. Proposals should be directed to the corresponding author and will undergo approval by the investigative team. To gain access after proposal approval, data requestors will need to sign a data access agreement. Data will be available for 1 year after proposal approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 12 months and ending 36 months following article publication.
Access Criteria: Researcher will provide a proposal to the corresponding author by email or written letter and the proposal will undergo approval by the investigative team. A data access agreement will be required.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blue Light | Amber Light | Ambient White Light
Started | 2 (The two participants that were enrolled in the study, withdrew between day 13 and 15 respectively due to symptoms of their cancer.) | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated due to slow recruitment. Participants enrolled only to the Blue Light Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blue Light | Amber Light | Ambient White Light | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (7.78) |  |  | 68.5 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 2 |  |  | 2
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Complete Response
Description: Rate of complete response to neoadjuvant chemoradiation upon restaging
Time Frame: Six months
Population: Trial was terminated before the outcome measure data were collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Sleep Quality
Description: The Pittsburgh Sleep Quality Index (PSQI) - seven component scores on scale 0-3 are summed for a total score: Lowest score: 0 (best sleep quality), Highest score: 21 (worst sleep quality).
Time Frame: Six months
Population: No data were collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Pain Control
Description: The Brief Pain Inventory (BPI) - Lowest score: 0 (lowest pain severity, least interference with function), Highest score: 10 (greatest pain severity, most interference with function).
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Quality of Life as Determined by WHO QOL Survey.
Description: The World Health Organization Quality of Life Brief Version - WHOQOL-Bref: scores calculated for each of four domains: physical, psychological, social, and environmental - Lowest score: 4 (very dissatisfied), Highest score: 20 (very satisfied).
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Functional Status
Description: The Karnofsky Performance Scale - Lowest score 0% (dead), Highest score 100% (normal; no complaints, no evidence of disease)
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Weight Loss
Description: Change in BMI will be used as a marker of nutritional status.
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Circadian Activation
Description: Rev-erb alpha concentration
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Immune Modulation
Description: Cytokine levels (IL-10,IL-6)
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Chemoradiation Tolerance
Description: Percentage of planned chemoradiation completed
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Prealbumin Level
Description: Change in prealbumin level will be used as a measure of nutritional status
Time Frame: Six months
Population: No data collected.
Arm/Group | Blue Light | Amber Light | Ambient White Light
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 15 days
Description: Study terminated due to slow recruitment. Participants enrolled only to the Blue Light Arm.
Arm/Group | Blue Light | Amber Light | Ambient White Light
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT06164691/Prot_SAP_000.pdf